CLINICAL TRIAL: NCT04903327
Title: Treatment of COVID-19-Induced Acute Respiratory Distress: A Phase 2 Study of Intravenous Administration of Allogeneic Adipose-Derived Mesenchymal Stem Cells
Brief Title: Study of Intravenous COVI-MSC for Treatment of COVID-19-Induced Acute Respiratory Distress
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to considerably slow enrollment, unable to reach enrollment targets
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSC-COV-201BR
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-MSC (Experimental): Subjects will receive intravenous infusions of COVI-MSC (two vials or a total of ≈ 30 million cells) on Day 0, Day 2, and Day 4
  Interventions: Biological: COVI-MSC
- Placebo (Placebo Comparator): Subjects will receive intravenous infusions of placebo (two vials) on Day 0, Day 2, and Day 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-MSC — COVI-MSC are allogeneic culture-expanded adipose-derived mesenchymal stem cells
  Arms: COVI-MSC
Drug: Placebo — Excipient solution
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized controlled study to assess the safety and efficacy of COVI-MSC in the setting of current standard of care treatments for COVID-19 infection in hospitalized subjects with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
This is a Phase 2 randomized controlled study to assess the safety and efficacy of COVI-MSC in the setting of current standard of care treatments for COVID-19 infection in hospitalized subjects with acute respiratory distress syndrome.

COVI-MSC or placebo will be administered intravenously on Day 0, Day 2, and Day 4.

Acceptable standard of care treatments for COVID-19 include all approved or emergency use authorized treatments for COVID-19, even if used off-label.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed SARS-CoV-2 infection as determined by an approved polymerase chain reaction (PCR) or an approved antigen test of any specimen
* Hospitalized with COVID-19-induced ARD or ARDS (any severity) with a PaO2/FiO2 (PF ratio) ≤ 300
* Requires oxygen supplementation at Screening
* Willing to follow contraception guidelines

Exclusion Criteria:

* Current standard of care treatments for COVID-19 appear to be working and the subject is clinically improving
* A previous stem cell infusion unrelated to this trial
* Certain medical conditions that pose a safety risk to the subject
* Pregnant or breast feeding or planning to during the study
* Suspected uncontrolled active bacterial, fungal, viral, or other infection
* History of splenectomy, lung transplant, or lung lobectomy
* Concurrent participation in another clinical trial involving therapeutic interventions
* Expected survival or time to withdrawal of life-sustaining treatments expected to be <7 days
* Has an existing "Do Not Intubate" order
* Has undergone home mechanical ventilation (noninvasive ventilation or via tracheotomy) expect for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rate at Day 28 | Baseline through Day 28
  All-cause mortality rate at Day 28

SECONDARY OUTCOMES:
All-cause mortality rate at Day 60 and Day 90 | Baseline through Day 60 and Day 90
  All-cause mortality rate at Day 60 and Day 90
Number of ventilator-free days through Day 28 | Baseline through Day 28
  Number of ventilator-free days through Day 28
Number of ICU days through Day 28 | Baseline through Day 28
  Number of ICU days through Day 28
Change in clinical status | Baseline to Day 28
  Change in clinical status as assessed using the 11-point WHO Clinical Progression Scale (0-10, where lower score means a better outcome)
Change in oxygenation | Baseline to Day 2, Day 4, Day 6, Day 14 and Day 28
  Change in oxygenation as assessed using PaO2:FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (6):
- Brazil (6):
  - Hospital São Rafael S.A. - Instituto D'Or de Pesquisa e Ensino, Salvador, Estado de Bahia
  - Santa Casa de Misericórdia da Bahia (Hospital Santa Izabel), Salvador, Estado de Bahia
  - Saraiva & Berlinger Ltda. - EPP (IPECC), Campinas, São Paulo
  - CECIP JAU - Centro de Estudos Clínicos do Interior Paulista Ltda., Jaú, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos Ltda. - EPP, São Bernardo do Campo, São Paulo
  - Impar Serviços Hospitalares S/A (Hospital Nove de Julho), São Paulo, São Paulo